CLINICAL TRIAL: NCT04513145
Title: Multimodal Periarticular Analgesic Injection With and Without Surgeon-Administered Adductor Canal Block During Total Knee Arthroplasty: A Randomized Controlled Trial
Brief Title: Adductor Canal Block
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: OrthoCarolina Research Institute, Inc. (Other)
Collaborators: Towson Orthopaedic Associates (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9172
Record Dates: First submitted 2020-08-11; First posted 2020-08-14 (Actual); Last update posted 2025-04-28 (Actual); Status verified 2025-04

CONDITIONS: Osteoarthritis; Total Knee Replacement
MeSH Terms: conditions — Osteoarthritis | interventions — Ropivacaine; Sodium Chloride; Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Both the investigator and participant will be blinded to the injection administered perioperatively
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment Group (Ropivacaine) (Experimental): The treatment group will consist of patients undergoing total knee arthroplasty who receive standardized 100 cc periarticularinjection into the lateral femoral periosteum, posterior capsule, medial periosteum, capsule and skin. Patients will then receive 10cc of ropivacaineinto their adductor canal.This will be administered by injecting into the adductor canal without dissecting down to the saphenous nerve and without ultrasound guidance.
  Interventions: Drug: Ropivacaine injection; Procedure: Total Knee Arthroplasty
- Control Group (Saline) (Placebo Comparator): The control group will consist of patients undergoing total knee arthroplasty who receive a standardized periarticular injection into the lateral femoral periosteum, posterior capsule, medial periosteum, capsule and skin. Patients randomized in this group will then receive 10cc of saline into their adductor canal. This will be administered by injecting into the adductor canal without dissecting down to the saphenous nerve and without ultrasound guidance.
  Interventions: Drug: Saline Injection; Procedure: Total Knee Arthroplasty

INTERVENTIONS:
Drug: Ropivacaine injection — Ropivacaine is a local anesthetic that is FDA approved for local anesthetic nerve block.
  Arms: Treatment Group (Ropivacaine)
Drug: Saline Injection — Saline will be used as a placebo injection
  Arms: Control Group (Saline)
Procedure: Total Knee Arthroplasty — All subjects participating in this study will undergo primary total knee arthroplasty

SUMMARY:
The investigators aim to investigate whether the addition of a surgeon-administered adductor canal blockade to a multimodal periarticular injection cocktail provides additional pain relief for patients undergoing total knee arthroplasty. This study will help identify the effectiveness of surgeon-administered adductor canal blockade in perioperative pain control for patients undergoing total knee arthroplasty

DETAILED DESCRIPTION:
Local anesthesia is an important component of multimodal pain management during the perioperative period for total knee arthroplasty, particularly with increased emphasis on early mobilization and decreased length of stay. Periarticular injections and regional nerve blocks are both effective in providing short-term pain relief when administered in isolation, and multiple randomized controlled trials have demonstrated that when administered in conjunction with one another, they also provide a synergistic effect.

Periarticular injections are the simplest mechanism for infiltrating the surgical site with analgesic medications, and these provide effective pain relief. One described technique involves infiltrating this mixture into the lateral femoral periosteum, posterior capsule, medial periosteum, capsule and skin during various portions of a total knee arthroplasty. This is the technique used in our practice.

Regional nerve blocks also have beneficial effects on pain, early mobilization and length of stay. Traditionally, anesthesiologist-administered femoral nerve blocks were utilized for this purpose. The femoral nerve consists of 4 main branches:the terminal portion of the vastusmedialis branch innervates the medial collateral ligament (MCL). The terminal portion of the vastusintermedius branch innervates the anterosuperior aspect of the knee capsule. The terminal portion of the vastuslateralis branch does not innervate the knee capsule. The saphenous nerve is the terminal sensory branch of the femoral nerve and travels in the adductor canal. It gives off an infrapatellar branch which exits the adductor canal to innervate the skin on the anteromedial aspect of the knee and the anteroinferior aspect of the knee capsule. Blockade of the entire femoral nerve results in significant quadriceps motor deficits.

Adductor canal blocks can be targeted to anesthetize only the saphenous branch of the femoral nerve, however, and this spares the motor innervation to the quadriceps. Multiple randomized controlled trials have shown that these adductor canal blockades provide equivalent analgesic effects to femoral nerve blocks without associated deficits in quadriceps strength. In one study, quadriceps strength was measured immediately prior to and immediately following placement of femoral and adductor can blocks in patients undergoing TKA. After the femoral block, quadriceps strength decreased to 16% of the baseline pre-block value. After the adductor-canal-block, however, strength increased to 193% of the pre-block value. MRI measurements, cadaveric injections, and dissections have shown that a surgeon-performed injection of the saphenous nerve from within the knee after it exits from the adductor canal is a feasible procedure, and a randomized controlled trial found that a surgeon-administered adductor canal blockade was non-inferior to the traditional adductor canal blockade administered by an anesthesiologist. This technique is simple and can be easily performed during administration of a periarticular injection. It is unclear based on the current literature whether this surgeon-administered adductor canal blockade provides a synergistic effect on pain relief when combined with a periarticular injection.

Treatment Group:

The treatment group will consist of patients undergoing total knee arthroplasty who receive standardized 100 cc periarticular injection into the lateral femoral periosteum, posterior capsule, medial periosteum, capsule and skin. Patients will then receive 10cc of ropivacaine into their adductor canal. This will be administered by injecting into the adductor canal without dissecting down to the saphenous nerve and without ultrasound guidance.

Comparison (Control) Group:

The control group will consist of patients undergoing total knee arthroplasty who receive a standardized periarticular injection into the lateral femoral periosteum, posterior capsule, medial periosteum, capsule and skin. Patients randomized in this group will then receive 10cc of saline into their adductor canal. This will be administered by injecting into the adductor canal without dissecting down to the saphenous nerve and without ultrasound guidance.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age 30-85undergoing first-time primary unilateral total knee arthroplasty for osteoarthritis and remaining hospitalized for at least one night

Exclusion Criteria:

1. Patients undergoing revision total knee arthroplasty
2. Patients undergoing bilateral total knee arthroplasty
3. Workers compensation patients
4. Patients undergoing total knee arthroplasty for post-traumatic arthritis
5. Patients with inflammatory arthritis
6. Patients with any previous surgery on the operative knee which involved an arthrotomy
7. Patients taking opioids prior to total knee arthroplasty
8. Patients with a known history of drug or alcohol abuse
9. Patients undergoing total knee arthroplasty at an ambulatory surgery center, or being discharged home from the hospital on the same day as their procedure (planned)
10. Patients who have had a total knee arthroplasty performed on the contralateral knee

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2020-10-09 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain, as defined by patient-reported NPRS pain scores on a scale of 0-10 on Postoperative day 1 | Approximately 24 hours following closure
  Pain will be measured before discharge on postoperative day 1 on a scale of 0 (no pain) - 10 (worst pain)

SECONDARY OUTCOMES:
Postoperative pain, as defined by patient-reported NPRS pain scores on a scale of 0-10 on Postoperative day 0, 1, 2, 4 and at 4-6 week postoperative visit | Every 6 hours for postoperative day 0-2, every 6 hours on postoperative day 4, and at 4-6 week visit
  Postoperative pain, as defined by patient-reported NPRS pain scores on a scale of 0 (no pain) - 10 (worst pain) on:
  * Postoperative day 0: in PACU and Q 6 hours
  * Postoperative day 1: Q 6 hours
  * Postoperative day 2: Q 6 hours via pain diary
  * Postoperative day 4: Q 6 hours via pain diary
  * 4-6 weeks postoperatively in office visit.
Timed Up & Go test | 24 hours following surgical closure
  Timed up & go test administered on postoperative day 1 by physical therapy
Gait Assessment | 24 hours following surgical closure
  Assessment using 2 Minute walk test, administered by physical therapy on postoperative day #1
Range of Motion | 24 hours following surgical closure
  Range of motion in knee flexion and extension on postoperative day 1 administered by physical therapy
Range of Motion | 4-6 weeks
  Range of motion in knee flexion and extension at 4-6 week visit administered by treating surgeon
Quadriceps Strength | 24 hours following surgical closure
  Quadriceps Strength (motor blockade) as demonstrated by ability to have active extension and perform a straight leg raise at Physical Therapy on postoperative day # 0 and postoperative day #1 prior to discharge.
Patient Satisfaction with Pain | 4-6 week visit
  Patient-reported satisfaction with pain control on a 10-point Likert scale where 10 is the highest satisfaction
Pain Diary | 7 days following surgical closure
  Patient-reported opioid consumption in morphine milliequivalents in first 7 days postoperatively as recorded in a pain diary

CONTACTS AND LOCATIONS:
Overall Officials: Bryan D Springer, MD, Principal Investigator — OrthoCarolina Research Institute, Inc.
Locations (1):
- OrthoCarolina Research Institute, OrthoCarolina, P.A., Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to currently make individual participant data available to other researchers